CLINICAL TRIAL: NCT05652959
Title: Real-world Performance and Safety of Cerviron® Medical Device in the Treatment of Various Types of Vaginitis
Brief Title: Real-world Performance and Safety of Cerviron® in the Treatment of Vaginitis
Status: Completed | Type: Observational
Sponsor: Perfect Care Distribution (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Other Study IDs: CYRONRW/01/2022
Record Dates: First submitted 2022-11-18; First posted 2022-12-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Vaginitis; Bacterial Vaginosis
Keywords: vulvovaginitis; vaginal discharge; vaginal pH
MeSH Terms: conditions — Vaginitis; Vaginosis, Bacterial; Vulvovaginitis; Vaginal Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Cerviron® — Cerviron® is a medical device manufactured by PFC Pharma Manufacturing SL formulated following the provisions of the European Regulation 2017/745 on Medical Devices. Cerviron® is an invasive medical device of short-term use classified under annex VIII of the European Regulation 2017/745 as class IIb according to Rule 21. Cerviron® has a complex composition consisting of three topical pharmaceutical products - hexylresorcinol, collagen and bismuth subgallate - and four phytotherapeutic extracts - Calendula officinalis, Hydrastis canadensis, Thymus vulgaris extract and Curcuma longa. The Instructions for use specify its field of use as adjuvant in the treatment of acute and chronic vulvovaginitis of mechanical etiology, caused by changes of vaginal pH and changes of the vaginal flora and of cervical lesions of mechanical origin.

SUMMARY:
Vaginitis is a broad term that includes a range of gynecological disorders characterized by infection of vaginal mucosa, inflammation of vulva and alteration of the normal vaginal microflora. The most prevalent is bacterial vaginosis, followed by other clinical entities such as candidiasis, trichomoniasis and non-specific vaginitis.

A collection of clinical data was conducted to assess the tolerability of Cerviron® ovules in the treatment and management of various types of vaginitis in clinical practice. A total of 111 women aged between 20 and 70 years were recruited, 71 of whom were treated with Cerviron® ovules as monotherapy and 40 who used Cerviron® ovules as supportive treatment in conjunction with antibiotic therapy. The aim of our study was to assess the relief in vaginal symptoms and changes in the normal vaginal pH level after 3 months of treatment with Cerviron® medical device in real-life clinical practice settings.

DETAILED DESCRIPTION:
This study was designed as real-world evidence study with the primary purpose to assess the performance and tolerance of Cerviron® ovules in the treatment and management of various types of vulvovaginitis. The study collected clinical data from 28 different specialized gynecology clinical facilities. The study was conducted between May 20, 2021 and August 31, 2021.

The primary objective of this study was to assess the tolerability of Cerviron® ovules in the treatment and management of various types of vulvovaginitis, but also to confirm its performance both on symptoms relief and as a user-friendly device. The secondary objective of this study was to assess the performance of the medical device by clinical exam and patients' degree of satisfaction. The study design consisted of 3 or 4 visits over 90 ± 3 days. Cerviron® ovules were applied intravaginally, once per day, on the first day after menstruation and for 15 days during 3 consecutive months.

Data of 111 women aged between 20 and 70 years were analyzed, 71 of whom were treated with Cerviron® ovules as monotherapy and 40 who used Cerviron® ovules as supportive treatment in conjunction with anti-infectious therapy.

The symptoms recorded in the medical charts were followed to determine the performance of the medical device during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult females with a diagnosis of infectious or non-infectious vaginitis and treated with Cerviron® with or without anti-infectious treatment for at least three months:
* Negative result for Gardnerella vaginalis, Candida albicans, Trichomonas vaginalis.

Exclusion Criteria:

* Subjects with diagnosed abnormal genital bleeding;
* Subject with vulvar, vaginal or cervical cancer;
* Subjects with other inflammatory gynecological conditions.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Vaginitis is a common problem for women of all ages.
Study Population: Women aged between 20 and 70 years were treated with Cerviron® ovules as monotherapy and Cerviron® ovules as supportive treatment in conjunction with the antibiotic therapy having specific symptoms such as leukorrhea, vaginal itching, pain and a feeling of tension, vaginal burning, erythema, abnormal odor of vaginal secretions, dysuria and dyspareunia.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Safety of the medical device | 3 months
  the number of possible adverse Number of reactions observed during the treatment

SECONDARY OUTCOMES:
Improvement in the vaginal discharge aspect | 3 months
  Presence/absence of abnormal/normal vaginal discharge
Improvement in the association of vaginal symptoms (burn and pain) | 3 months
  Presence/absence of vaginal symptoms (burn and pain)
Improvement in vaginal irritation | 3 months
  Presence/absence of vaginal irritation
Measurement of vaginal pH | 3 months
  Normalization of vaginal pH values

CONTACTS AND LOCATIONS:
Overall Officials: Ema Peta, Study Director — Perfect Care Distribution
Locations (10):
- Romania (10):
  - Spitalul Clinic Dr. Ion Cantacuzino Bucharest, Bucharest
  - Med Life Humanitas Cluj-Napoca, Cluj-Napoca
  - Cabinet Medical - Dr. Saleh K. Majed, Craiova
  - Cabinet Medical - Dr. Surpanelu Oana, Iași
  - Clinica Natisan Pitesti, Piteşti
  - Cabinet Dr. Rădulescu G. Mihaela Elena, Râmnicu Vâlcea
  - Pan Medical Sibiu, Sibiu
  - Cabinet Dr. Ioana Trotea Targu Jiu, Târgu Jiu
  - Clinica Medicala Dr. Cioata Ionel Trifon, Timișoara
  - Spitalul Judetean de Urgenta Tulcea, Tulcea

REFERENCES:
- [Background] Hainer BL, Gibson MV. Vaginitis. Am Fam Physician. 2011 Apr 1;83(7):807-15. PMID 21524046
- [Background] Saraf VS, Sheikh SA, Ahmad A, Gillevet PM, Bokhari H, Javed S. Vaginal microbiome: normalcy vs dysbiosis. Arch Microbiol. 2021 Sep;203(7):3793-3802. doi: 10.1007/s00203-021-02414-3. Epub 2021 Jun 13. PMID 34120200
- [Background] Verstraelen H, Verhelst R, Vaneechoutte M, Temmerman M. Group A streptococcal vaginitis: an unrecognized cause of vaginal symptoms in adult women. Arch Gynecol Obstet. 2011 Jul;284(1):95-8. doi: 10.1007/s00404-011-1861-6. Epub 2011 Feb 19. PMID 21336834
- [Background] Coudray MS, Madhivanan P. Bacterial vaginosis-A brief synopsis of the literature. Eur J Obstet Gynecol Reprod Biol. 2020 Feb;245:143-148. doi: 10.1016/j.ejogrb.2019.12.035. Epub 2019 Dec 24. PMID 31901667
- [Background] Owen MK, Clenney TL. Management of vaginitis. Am Fam Physician. 2004 Dec 1;70(11):2125-32. PMID 15606061
- [Background] Brown H, Drexler M. Improving the Diagnosis of Vulvovaginitis: Perspectives to Align Practice, Guidelines, and Awareness. Popul Health Manag. 2020 Oct;23(S1):S3-S12. doi: 10.1089/pop.2020.0265. PMID 32997581